CLINICAL TRIAL: NCT02562235
Title: Open-label, Individual Dose Titration Study to Evaluate Safety, Tolerability and Pharmacokinetics of Riociguat in Children From 6 to Less Than 18 Years of Age With Pulmonary Arterial Hypertension (PAH)
Brief Title: Riociguat in Children With Pulmonary Arterial Hypertension (PAH)
Acronym: PATENT-CHILD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15681; 2014-003952-29 (EudraCT Number)
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary arterial hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Riociguat (Experimental): Participants with age ≥6 to <18 years received riociguat up to 2.5 mg three times a day (titration between 1.0 mg and 2.5 mg) for up to 8 weeks during the individual dose titration (IDT) phase, and followed with the last dose administered in the IDT phase for up to 16 weeks during the maintenance phase. Down-titration (up to 0.5 mg) of the dose for safety reasons was allowed at any time.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — For children with body-weight <50 kg at screening: body-weight adjusted dose equivalent to the exposure of (0.5 mg) 1.0 - 2.5 mg three times a day, IDT in adults treated for PAH; oral suspension. For children ≥50 kg at screening: 1.0 to 2.5 mg three times a day; oral tablet.

SUMMARY:
This study was designed to evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of riociguat at age-, sex- and body-weight-adjusted doses of 0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg and 2.5 mg TID in children from ≥6 to less than 18 years with pulmonary arterial hypertension (PAH) group 1. The study design consisted of a main study part followed by an optional long-term extension part. The main treatment period consisted of two phases: titration phase up to 8 weeks and a maintenance phase up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 years to less than 18 years of age with pulmonary arterial hypertension (PAH)
* Diagnosed with PAH :

  * Idiopathic (IPAH)
  * Hereditable (HPAH)
  * PAH associated with (APAH)

    * Connective tissue disease
    * Congenital heart disease with shunt closure more than 6 months ago (no open shunts, confirmed by RHC no less than 4 months after surgery)

Regardless of the type of PAH, the following findings are not exclusionary:

--- Patent foramen ovale (PFO) and asymptomatic, isolated, ostium secundum atrial septal defect (OS-ASD) ≤ 1 cm (both confirmed by echocardiogram) and not associated with hemodynamic alterations indicative of significant shunt, e.g. Qp/Qs ratio less <1.5:1 are not exclusionary

* PAH diagnosed by right heart catheterization (RHC) at any time prior to enrolment (for patients with closed shunts - RHC no less than 4 months after surgery)
* PAH confirmed by a RHC at any time prior to start of study, with mean pulmonary artery pressure (PAPmean) ≥25 mmHg at rest, pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure (LVEDP) ≤15 mmHg, and pulmonary vascular resistance (PVR) >240 dyn•sec•cm^-5 (i.e., ≥3.0 wood units•m^2)
* Patients must be on standard of care PAH medications, allowing Endothelin Receptor Antagonists (ERA) and/or Prostacyclin Analogues (PCA), for at least 12 weeks prior to baseline visit.

Two groups of patients will be included:

* Prevalent: Patients currently on PAH medication (allowing ERA and/or PCA) who need additional treatment (discretion of the investigator)
* Incident: Treatment naïve patients initiated on PAH medication (allowing ERA and /or PCA) and then riociguat added once patients are stable on standard of care

  * WHO functional class I-III
  * Adolescent females of childbearing potential can only be included in the study if a pregnancy test is negative. Adolescent females of childbearing potential must agree to receive sexual counseling and use effective contraception as applicable. 'Effective contraception' is defined as progestogen-only hormonal contraception associated with inhibition of ovulation (implant), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), or any combination of adequate methods of birth control (e.g. condoms with hormonal contraception). Agreement to use contraception is required from the signing of the informed consent form up until 4 weeks after the last study drug administration.
  * Young men must agree to use adequate contraception when sexually active.
  * Written inform consent provided and if applicable child assent provided

Exclusion Criteria:

* Concomitant use of the following medications: phosphodiesterase (PDE) 5 inhibitors (such as sildenafil, tadalafil, vardenafil) and non-specific phosphodiesterase (PDE) inhibitors (theophylline, dipyridamole), nitrates or NO donors (such as amyl nitrite) in any form

  -- Pretreatment with NO donors (e.g. nitrates) within the last 2-weeks before visit 1. The use of any drug including NO acutely for testing during catheterization is not an exclusion criterion.
* Active state of hemoptysis or pulmonary hemorrhage, including those events managed by bronchial artery embolization or any history of bronchial artery embolization or massive hemoptysis within 3 months prior to screening
* Systolic blood pressure (SBP) more than 5 mmHg lower than the age-, sex- and height-adapted level of the 50th SBP percentile (NHBPEP, 2004)
* History of left-sided heart disease, including valvular disease or heart failure
* Pulmonary hypertension related to conditions other than specified in the inclusion criteria
* WHO functional class IV
* Pulmonary veno-occlusive disease
* Screening aspartate transaminase (AST) and/ or alanine transaminase (ALT) more than 3 times the upper limit of normal (ULN)
* Severe restrictive lung disease
* Severe congenital abnormalities of the lung, thorax, and diaphragm
* Clinically relevant hepatic dysfunction (especially Child Pugh C)
* Renal insufficiency (estimated glomerular filtration rate <30 mL/min/1.73m^2 e.g. calculated based on Schwartz formula)
* PH associated with idiopathic interstitial pneumonia (PH-IIP)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2027-08-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- Clínica Imbanaco S.A.S, Cali, Valle del Cauca Department, Colombia
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Deutsches Herzzentrum der Charité (DHZC), Berlin
- Hungary (2):
  - Gottsegen Gyorgy Orszagos Kardiovaszkularis Intezet, Budapest
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
- Azienda Ospedale-Università di Padova - UOC Cardiologia Pediatrica, Padua, Veneto, Italy
- Japan (4):
  - Aichi Children's Health and Medical Center, Ōbu, Aichi-ken
  - The University of Osaka Hospital, Suita, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Keio University Hospital, Shinjuku-ku, Tokyo
- Mexico (2):
  - Instituto Nacional de Cardiología "Ignacio Chávez", México D.F., Mexico City
  - Operadora de Hospitales Angeles S. A. de C. V., Huixquilucan
- Wojewodzki Szpital Specjalistyczny - Wroclaw, Wroclaw, Poland
- Veterans General Hospital, Kaohsiung City, Taiwan
- Hacettepe Universitesi Tip Fakultesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 9 countries or regions between 29-Oct-2015 (first participant first visit) and 07-Mar-2020 (last participant last visit of main study part). The long-term extension part of the study is ongoing.
Pre-assignment Details: A total of 26 participants were screened. Of them, 2 participants were screening failures and 24 participants received study treatment.
Groups:
- Riociguat >=6 to <18 Years: Participants with age ≥6 to <18 years received riociguat up to 2.5 mg three times a day (titration between 1.0 mg and 2.5 mg) for up to 8 weeks during the individual dose titration (IDT) phase, and followed with the last dose administered in the IDT phase for up to 16 weeks during the maintenance phase. Down-titration (up to 0.5 mg) of the dose for safety reasons was allowed at any time.
Period: Overall Study
Arm/Group | Riociguat >=6 to <18 Years
Started | 24
Completed | 21
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): All participants who were assigned to receive study medication and had received at least one dose of the study medication.
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (2.8) [lower limit 2.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not reported | 24
Bone age compared to chronological age [Count of Participants; unit: Participants] — X-ray of left hand was performed for each participant and bone age was determined centrally by a specialist. For each participant, bone age was compared to chronological age and assessed as as "delayed, in accordance or advanced".
  Participants
    Delayed | 1
    In accordance | 12
    Advanced | 10
    Missing | 1
WHO functional class [Count of Participants; unit: Participants] — The World Health Organization (WHO) functional class describes how severe a patient's pulmonary hypertension (PH) symptoms are. There are four different classes - I is the mildest and IV the most severe form of PH.
  Participants
    Class I | 1
    Class II | 18
    Class III | 5
    Class IV | 0
Heart rate [Mean (Standard Deviation); unit: Beats per minute (BPM)] | 84.5 (19.0) [lower limit 19.0]
Diastolic blood pressure [Mean (Standard Deviation); unit: millimetre of mercury (mmHg)] | 63.8 (7.9) [lower limit 7.9]
Systolic blood pressure [Mean (Standard Deviation); unit: millimetre of mercury (mmHg)] | 112.9 (10.9) [lower limit 10.9]
Respiratory Rate [Mean (Standard Deviation); unit: Breath per minute] — Population: Participants in SAF with evaluable data for this measurement
  Breath per minute
    number analyzed (Participants) | 21
    (all) | 19.6 (4.4)
6-minute walking distance [Mean (Standard Deviation); unit: Meter] — 6-minute walking distance (6MWD) is a exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. An increase in the distance walked indicates improvement in basic mobility. Population: Participants in SAF with evaluable data for this measurement
  Meter
    number analyzed (Participants) | 23
    (all) | 442.12 (109.67)
N-terminal prohormone brain-type natriuretic peptide [Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)] — Laboratory biomarkers N-terminal prohormone brain-type natriuretic peptide (NT-proBNP) or brain-type natriuretic peptide (BNP) were tested for the participants. When both tests were available, NT-proBNP was chosen over BNP and the same test was performed at every required visit. Population: Participants in SAF with evaluable data for this measurement
  Picograms per milliliter (pg/mL)
    number analyzed (Participants) | 15
    (all) | 982.68 (1595.77)
Brain-type natriuretic peptide [Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)] — Laboratory biomarkers N-terminal prohormone brain-type natriuretic peptide (NT-proBNP) or brain-type natriuretic peptide (BNP) were tested for the participants. When both tests were available, NT-proBNP was chosen over BNP and the same test was performed at every required visit. Population: Participants in SAF with evaluable data for this measurement
  Picograms per milliliter (pg/mL)
    number analyzed (Participants) | 7
    (all) | 10.46 (9.10)
Quality of life evaluated by SF-10 questionnaire physical summary score [Mean (Standard Deviation); unit: Scores on a scale] — SF-10 is a parent-completed health survey for children that contains 10 questions adapted from the Child Health Questionnaire. It is scored using nom-based scoring to produce physical and psychosocial health summary measures. The possible range for the physical measure is -10.9 to 57.2 scores and higher scores indicate more favorable functioning.
  Scores on a scale | 30.964 (13.335) [lower limit 13.335]
Quality of life evaluated by SF-10 questionnaire psychosocial summary score [Mean (Standard Deviation); unit: Scores on a scale] — SF-10 is a parent-completed health survey for children that contains 10 questions adapted from the Child Health Questionnaire. It is scored using nom-based scoring to produce physical and psychosocial health summary measures. The possible range for the psychosocial measure is 8.8 to 62.3 scores and higher scores indicate more favorable functioning.
  Scores on a scale | 48.765 (8.263) [lower limit 8.263]
Quality of life evaluated by PedsQL total scale score [Mean (Standard Deviation); unit: Scores on a scale] — PedsQL Generic Core Scales were designed to measure health-related quality of life in children and adolescents. It has 4 dimensions: physical functioning, emotional functioning, social functioning and school functioning. 3 Summary Scores of PedsQL were calculated from the scales including total scale score, physical health summary score (physical functioning) and psychosocial health summary score (emotional, social and school functioning). Responses of the questions are transformed to a 0-100 scale. Higher scores indicate better quality of life. Population: Participants in SAF with evaluable data for this measurement
  Scores on a scale
    number analyzed (Participants) | 21
    (all) | 69.77 (16.29)
Quality of life evaluated by PedsQL physical health summary score [Mean (Standard Deviation); unit: Scores on a scale] — PedsQL Generic Core Scales were designed to measure health-related quality of life in children and adolescents. It has 4 dimensions: physical functioning, emotional functioning, social functioning and school functioning. 3 Summary Scores of PedsQL were calculated from the scales including total scale score, physical health summary score (physical functioning) and psychosocial health summary score (emotional, social and school functioning). Responses of the questions are transformed to a 0-100 scale. Higher scores indicate better quality of life. Population: Participants in SAF with evaluable data for this measurement
  Scores on a scale
    number analyzed (Participants) | 21
    (all) | 64.43 (15.80)
Quality of life evaluated by PedsQL psychosocial health summary score [Mean (Standard Deviation); unit: Scores on a scale] — PedsQL Generic Core Scales were designed to PedsQL Generic Core Scales were designed to measure health-related quality of life in children and adolescents. It has 4 dimensions: physical functioning, emotional functioning, social functioning and school functioning. 3 Summary Scores of PedsQL were calculated from the scales including total scale score, physical health summary score (physical functioning) and psychosocial health summary score (emotional, social and school functioning). Responses of the questions are transformed to a 0-100 scale. Higher scores indicate better quality of life. Population: Participants in SAF with evaluable data for this measurement
  Scores on a scale
    number analyzed (Participants) | 21
    (all) | 72.62 (19.20)
Estimate right atrial pressure [Mean (Standard Deviation); unit: millimetre of mercury (mmHg)] — Estimate right atrial pressure was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  millimetre of mercury (mmHg)
    number analyzed (Participants) | 18
    (all) | 9.2 (2.9)
Left ventricular eccentricity index [Mean (Standard Deviation); unit: Ratio] — Left ventricular (LV) eccentricity index (EI) is defined as the ratio of the LV long axis to the LV transverse diameter, measured at end systole and end diastole by echocardiography. The value of EI > 1.0 is abnormal and suggests right ventricle (RV) overload. Population: Participants in SAF with evaluable data for this measurement
  Ratio
    number analyzed (Participants) | 17
    (all) | 2.099 (1.275)
Pulmonary artery acceleration time [Mean (Standard Deviation); unit: Millisecond (msec)] — Pulmonary artery acceleration time was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  Millisecond (msec)
    number analyzed (Participants) | 17
    (all) | 91.568 (36.853)
Right ventricular cardiac index [Mean (Standard Deviation); unit: Liter/minute/square meter (L/min/m^2)] — Right ventricle (RV) cardiac index (CI) was measured by echocardiography and calculated by dividing the cardiac output (stroke volume × heart rate) by the body surface area. The change in RV CI should not be understood solely but associated with other conditions of the participants. Population: Participants in SAF with evaluable data for this measurement
  Liter/minute/square meter (L/min/m^2)
    number analyzed (Participants) | 16
    (all) | 4.343 (1.599)
Right ventricular cardiac output [Mean (Standard Deviation); unit: Liter per minute (L/min)] — Right ventricular cardiac output was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  Liter per minute (L/min)
    number analyzed (Participants) | 16
    (all) | 5.511 (2.093)
Right atrial diastolic area [Mean (Standard Deviation); unit: Square centimeter (cm^2)] — Right atrial diastolic area was measured by echocardiography. Number of subjects with right atrial diastolic area data at baseline: n=18 Population: Participants in SAF with evaluable data for this measurement
  Square centimeter (cm^2)
    number analyzed (Participants) | 18
    (all) | 16.944 (11.071)
Right atrial diastolic area index [Mean (Standard Deviation); unit: Ratio] — Right atrial (RA) diastolic area index was measured by echocardiography and calculated by dividing the RA area at end-diastole by the body surface area. The RA area index is a reflection of RA volume at end-diastole. The change in the index should not be understood solely but associated with other conditions of the participants. Population: Participants in SAF with evaluable data for this measurement
  Ratio
    number analyzed (Participants) | 18
    (all) | 12.788 (6.977)
Right atrial systolic area [Mean (Standard Deviation); unit: Square centimeter (cm^2)] — Right atrial systolic area was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  Square centimeter (cm^2)
    number analyzed (Participants) | 18
    (all) | 12.017 (9.391)
Right atrial systolic area index [Mean (Standard Deviation); unit: Ratio] — Right atrial (RA) systolic area index was measured by echocardiography and calculated by dividing the RA area at end-systole by the body surface area. The RA area index is a reflection of RA volume at end-systole. The change in the index should not be understood solely but associated with other conditions of the participants. Population: Participants in SAF with evaluable data for this measurement
  Ratio
    number analyzed (Participants) | 18
    (all) | 8.996 (6.021)
Right ventricular fractional area change [Mean (Standard Deviation); unit: Percentage (%)] — Right ventricular fractional area change was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  Percentage (%)
    number analyzed (Participants) | 17
    (all) | 25.7 (8.5)
Right ventricular diastolic area [Mean (Standard Deviation); unit: Square centimeter (cm^2)] — Right ventricular diastolic area was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  Square centimeter (cm^2)
    number analyzed (Participants) | 17
    (all) | 27.155 (11.993)
Right ventricular diastolic area index [Mean (Standard Deviation); unit: Ratio] — Right ventricular (RV) diastolic area index was measured by echocardiography and calculated by dividing the RV area at end-diastole by the body surface area. The RV area index is a reflection of RV volume at end-diastole. The change in the index should not be understood solely but associated with other conditions of the participants. Population: Participants in SAF with evaluable data for this measurement
  Ratio
    number analyzed (Participants) | 17
    (all) | 20.722 (6.564)
Right ventricular systolic area [Mean (Standard Deviation); unit: Square centimeter (cm^2)] — Right ventricular systolic area was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  Square centimeter (cm^2)
    number analyzed (Participants) | 17
    (all) | 20.235 (9.343)
Right ventricular systolic area index [Mean (Standard Deviation); unit: Ratio] — Right ventricular (RV) systolic area index was measured by echocardiography and calculated by dividing the RV area at end-systole by the body surface area. The RV area index is a reflection of RV volume at end-systole. The change in the index should not be understood solely but associated with other conditions of the participants. Population: Participants in SAF with evaluable data for this measurement
  Ratio
    number analyzed (Participants) | 17
    (all) | 15.613 (5.745)
Systolic pulmonary artery pressure [Mean (Standard Deviation); unit: millimetre of mercury (mmHg)] — Systolic pulmonary artery pressure was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  millimetre of mercury (mmHg)
    number analyzed (Participants) | 6
    (all) | 117.2 (51.6)
Tricuspid annular plane systolic excursion [Mean (Standard Deviation); unit: Millimeter (mm)] — Tricuspid annular plane systolic excursion was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  Millimeter (mm)
    number analyzed (Participants) | 17
    (all) | 18.82 (4.21)
Tricuspid regurgitation peak velocity [Mean (Standard Deviation); unit: Meter/second (m/s)] — Tricuspid regurgitation peak velocity was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  Meter/second (m/s)
    number analyzed (Participants) | 11
    (all) | 4.915 (1.100)
Pericardial effusion [Mean (Standard Deviation); unit: Millimeter (mm)] — Pericardial effusion was measured by echocardiography. Population: Participants in SAF with evaluable data for this measurement
  Millimeter (mm)
    number analyzed (Participants) | 2
    (all) | 1.280 (0.212)
Platelets [Mean (Standard Deviation); unit: Giga platelets per liter] — Hematology parameters were collected and analyzed.
  Giga platelets per liter | 218.8 (50.6) [lower limit 50.6]
Lymphocytes/leucocytes ratio [Mean (Standard Deviation); unit: Percentage of leucocytes in blood] — Hematology parameters were collected and analyzed.
  Percentage of leucocytes in blood | 48.98 (8.15) [lower limit 8.15]
Neutrophils/leucocytes ratio [Mean (Standard Deviation); unit: Percentage of leucocytes in blood] — Hematology parameters were collected and analyzed.
  Percentage of leucocytes in blood | 18.71 (10.37) [lower limit 10.37]
Alanine aminotransferase [Mean (Standard Deviation); unit: Units per liter (U/L)] — Clinical chemistry parameters were collected and analyzed.
  Units per liter (U/L) | 18.71 (10.37) [lower limit 10.37]
Aspartate aminotransferase [Mean (Standard Deviation); unit: Units per liter (U/L)] — Clinical chemistry parameters were collected and analyzed.
  Units per liter (U/L) | 23.76 (8.38) [lower limit 8.38]
Urea [Mean (Standard Deviation); unit: microgram per deciliter (mg/dL)] — Clinical chemistry parameters were collected and analyzed. Population: Participants in SAF with evaluable data for this measurement
  microgram per deciliter (mg/dL)
    number analyzed (Participants) | 11
    (all) | 25.17 (7.23)
Gamma glutamyl transferase [Mean (Standard Deviation); unit: Units per liter (U/L)] — Clinical chemistry parameters were collected and analyzed. Population: Participants in SAF with evaluable data for this measurement
  Units per liter (U/L)
    number analyzed (Participants) | 20
    (all) | 16.9 (14.5)
Blood urea nitrogen [Mean (Standard Deviation); unit: microgram per deciliter (mg/dL)] — Clinical chemistry parameters were collected and analyzed. Population: Participants in SAF with evaluable data for this measurement
  microgram per deciliter (mg/dL)
    number analyzed (Participants) | 17
    (all) | 11.8 (4.7)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: milliliter/minute/1.73 square meter] — Clinical chemistry parameters were collected and analyzed.
  milliliter/minute/1.73 square meter | 117.877 (30.649) [lower limit 30.649]
Sodium [Mean (Standard Deviation); unit: millimole per Liter (mmol/L)] — Clinical chemistry parameters were collected and analyzed. Population: Participants in SAF with evaluable data for this measurement
  millimole per Liter (mmol/L)
    number analyzed (Participants) | 22
    (all) | 140.5 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events
Description: An adverse event (AE), including AE in relation to a medical device (i.e. Raumedic dosing pipette), is any untoward medical occurrence in a participant administered with a pharmaceutical product and does not necessarily have to have a causal relationship with this treatment. A serious AE (SAE) is any untoward medical occurrence that at any dose is resulting in death, is lifethreatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity. AEs occurring between start of study drug and up to 2 days after the last dose were defined as treatment-emergent AEs (TEAEs).
Time Frame: From start of study drug up to 2 days after the last dose of study drug in the main study part, up to 24 weeks plus/minus 5 days.
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 24
Participants
  Any TEAE | 20
  Any serious TEAE | 4

2. Primary Outcome: Change in Heart Rate From Baseline
Description: Mean change in heart rate from baseline is reported.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 21
Beats per minute (BPM) | 4.1 (10.1) [lower limit 10.1]

3. Primary Outcome: Change in Blood Pressure From Baseline
Description: Mean changes in systolic blood pressure (SBP) and diastolic blood pressure (DBP) from baseline are reported.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 21
millimetre of mercury (mmHg)
  SBP | -3.1 (10.5) [lower limit 10.5]
  DBP | -2.4 (10.0) [lower limit 10.0]

4. Primary Outcome: Change in Respiratory Rate From Baseline
Description: Mean change in respiratory rate from baseline is reported.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Breath per minute
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 18
Breath per minute | 0.3 (3.3) [lower limit 3.3]

5. Primary Outcome: Number of Subjects With Transitions From Baseline in Bone Age Compared to Chronological Age
Description: X-ray of left hand was performed for each participant and bone age was determined centrally by a specialist. For each participant, the bone age was compared to the chronological age and assigned to one of the categories - "delayed", "in accordance" or "advanced", indicating the advancement or delay in the growth of the bone. Number of participants who transitioned to another category different from baseline was calculated and is reported.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 21
Participants
  Transitioned from Delayed to In Accordance | 0
  Transitioned from Delayed to Advanced | 0
  Transitioned from In Accordance to Delayed | 1
  Transitioned from In Accordance to Advanced | 3
  Transitioned from In Accordance to Missing | 1
  Transitioned from Advanced to Delayed | 1
  Transitioned from Advanced to In Accordance | 0

6. Primary Outcome: Change in Hematology Parameters (Platelets) From Baseline
Description: Hematology parameters were collected. Parameters with a decrease or increase in the mean value compared to baseline are reported in this data set.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Giga platelets per Liter
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 20
Giga platelets per Liter | -4.4 (51.1) [lower limit 51.1]

7. Primary Outcome: Change in Hematology Parameters (Lymphocytes/Leucocytes Ratio) From Baseline
Description: as for outcome 6
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Percentage of leucocytes in blood
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 20
Percentage of leucocytes in blood | -4.77 (11.08) [lower limit 11.08]

8. Primary Outcome: Change in Hematology Parameter (Neutrophils/Leucocytes Ratio) From Baseline
Description: as for outcome 6
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Percentage of leucocytes in blood
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 20
Percentage of leucocytes in blood | 5.71 (11.73) [lower limit 11.73]

9. Primary Outcome: Change in Clinical Chemistry (Alanine Aminotransferase) From Baseline
Description: Clinical chemistry parameters were collected and analyzed. Parameters with a trend to lower or higher mean values from baseline are reported in this data set.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 21
Units per liter (U/L) | -1.01 (9.86) [lower limit 9.86]

10. Primary Outcome: Change in Clinical Chemistry (Aspartate Aminotransferase) From Baseline
Description: as for outcome 9
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 21
Units per liter (U/L) | -1.94 (6.52) [lower limit 6.52]

11. Primary Outcome: Change in Clinical Chemistry (Sodium) From Baseline
Description: as for outcome 9
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 19
millimole per Liter (mmol/L) | -1.0 (1.9) [lower limit 1.9]

12. Primary Outcome: Change in Clinical Chemistry (Blood Urea Nitrogen) From Baseline
Description: as for outcome 9
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: microgram per deciliter (mg/dL)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 14
microgram per deciliter (mg/dL) | 1.3 (4.3) [lower limit 4.3]

13. Primary Outcome: Change in Clinical Chemistry (eGFR) From Baseline
Description: Clinical chemistry parameters were collected and analyzed. Parameters with a trend to lower or higher mean values from baseline are reported in this data set. eGFR = estimated glomerular filtration rate
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: milliliter/minute/1.73 square meter
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 21
milliliter/minute/1.73 square meter | -4.459 (25.686) [lower limit 25.686]

14. Primary Outcome: Change in Clinical Chemistry (Urea) From Baseline
Description: as for outcome 9
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: microgram per deciliter (mg/dL)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 9
microgram per deciliter (mg/dL) | 4.06 (10.52) [lower limit 10.52]

15. Primary Outcome: Change in Clinical Chemistry (Gamma Glutamyl Transferase) From Baseline
Description: as for outcome 9
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 18
Units per liter (U/L) | 1.7 (4.0) [lower limit 4.0]

16. Primary Outcome: Plasma Concentration of Riociguat at Week 0
Description: For each participant, one blood sample was collected at one given time point. Values below lower limit of quantification (LLOQ) were substituted by 1/2 LLOQ for the calculation in statistics. Means at any time were only calculated if at least 2/3 of the individual data were measured and were above the limit of quantification (LOQ). Geometric mean and percentage geometric coefficient of variation (%CV) are reported. W = Week.
Time Frame: Week 0 (30-90 minutes post-dose; 2.5-4 hours post-dose)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Groups:
- Riociguat 1.0 mg or Equivalent - PK: Participants who received riociguat at 1.0 mg or body weight-adjusted dose equivalent to the exposure of 1.0 mg dose in adults at the day of PK measurement
Arm/Group | Riociguat 1.0 mg or Equivalent - PK
Number analyzed (Participants) | 22
microgram per liter (mcg/L)
  W0 (30-90 min post-dose) | 15.340 (90.536)
  W0 (2.5-4 h post-dose) | 17.791 (55.690)

17. Primary Outcome: Plasma Concentration of Riociguat at Week 4
Description: For each participant, one blood sample was collected at one given time point. Values below lower limit of quantification (LLOQ) were substituted by 1/2 LLOQ for the calculation in statistics. Means at any time were only calculated if at least 2/3 of the individual data were measured and were above the limit of quantification (LOQ). Geometric mean and percentage geometric coefficient of variation (%CV) are reported.
Time Frame: Week 4 (pre-dose)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Groups:
- Riociguat 0.5 mg or Equivalent - PK: Participants who received riociguat at 0.5 mg or body weight-adjusted dose equivalent to the exposure of 0.5 mg dose in adults at the day of PK measurement
- Riociguat 2.0 mg or Equivalent - PK: Participants who received riociguat at 2.0 mg or body weight-adjusted dose equivalent to the exposure of 2.0 mg dose in adults at the day of PK measurement
Arm/Group | Riociguat 0.5 mg or Equivalent - PK | Riociguat 1.0 mg or Equivalent - PK | Riociguat 2.0 mg or Equivalent - PK
Number analyzed (Participants) | 1 | 2 | 17
microgram per liter (mcg/L) | 4.510 (NA) — Value was not calculated due to very low number of participants. | 65.585 (47.727) | 31.126 (89.790)

18. Primary Outcome: Plasma Concentration of Riociguat at Week 8
Description: as for outcome 17
Time Frame: Week 8 (pre-dose)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Groups:
- Riociguat 2.5 mg or Equivalent - PK: Participants who received riociguat at 2.5 mg or body weight-adjusted dose equivalent to the exposure of 2.5 mg dose in adults at the day of PK measurement
Arm/Group | Riociguat 0.5 mg or Equivalent - PK | Riociguat 1.0 mg or Equivalent - PK | Riociguat 2.0 mg or Equivalent - PK | Riociguat 2.5 mg or Equivalent - PK
Number analyzed (Participants) | 2 | 1 | 1 | 15
microgram per liter (mcg/L) | 11.650 (244.238) | 27.100 (NA) — Value was not calculated due to very low number of participants. | 14.000 (NA) — Value was not calculated due to very low number of participants. | 32.381 (137.719)

19. Primary Outcome: Plasma Concentration of BAY60-4552 at Week 0
Description: BAY60-4552 is riociguat's active metabolite. For each participant, one blood sample was collected at one given time point and in that sample both riociguat and BAY60-4552 were measured. Values below lower limit of quantification (LLOQ) were substituted by 1/2 LLOQ for the calculation in statistics. Means at any time were only calculated if at least 2/3 of the individual data were measured and were above the limit of quantification (LOQ). Geometric mean and percentage geometric coefficient of variation (%CV) are reported. W = Week
Time Frame: Week 0 (30-90 minutes post-dose; 2.5-4 hours post-dose)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Arm/Group | Riociguat 1.0 mg or Equivalent - PK
Number analyzed (Participants) | 22
microgram per liter (mcg/L)
  W0 (30-90 min post-dose) | NA (NA) — Value was not calculated due to very low number of participants.
  W0 (2.5-4 h post-dose) | 3.922 (94.399)

20. Primary Outcome: Plasma Concentration of BAY60-4552 at Week 4
Description: BAY60-4552 is riociguat's active metabolite. For each participant, one blood sample was collected at one given time point and in that sample both riociguat and BAY60-4552 were measured. Values below lower limit of quantification (LLOQ) were substituted by 1/2 LLOQ for the calculation in statistics. Means at any time were only calculated if at least 2/3 of the individual data were measured and were above the limit of quantification (LOQ). Geometric mean and percentage geometric coefficient of variation (%CV) are reported.
Time Frame: Week 4 (pre-dose)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Arm/Group | Riociguat 0.5 mg or Equivalent - PK | Riociguat 1.0 mg or Equivalent - PK | Riociguat 2.0 mg or Equivalent - PK
Number analyzed (Participants) | 1 | 2 | 17
microgram per liter (mcg/L) | 12.700 (NA) — Value was not calculated due to very low number of participants. | 48.822 (193.584) | 38.579 (27.242)

21. Primary Outcome: Plasma Concentration of BAY60-4552 at Week 8
Description: as for outcome 20
Time Frame: Week 8 (pre-dose)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Arm/Group | Riociguat 0.5 mg or Equivalent - PK | Riociguat 1.0 mg or Equivalent - PK | Riociguat 2.0 mg or Equivalent - PK | Riociguat 2.5 mg or Equivalent - PK
Number analyzed (Participants) | 2 | 1 | 1 | 15
microgram per liter (mcg/L) | 23.065 (91.296) | 13.200 (NA) — Value was not calculated due to very low number of participants. | 49.600 (NA) — Value was not calculated due to very low number of participants. | 65.849 (26.864)

22. Secondary Outcome: Change in 6-minute Walking Distance From Baseline
Description: 6-minute walking distance (6MWD) is a exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. An increase in the distance walked indicates improvement in basic mobility.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 19
Meter | 23.01 (68.80) [lower limit 68.80]

23. Secondary Outcome: Number of Subjects With Change in WHO Functional Class From Baseline
Description: The World Health Organization (WHO) functional class describes how severe a patient's pulmonary hypertension (PH) symptoms are. There are four different classes - I is the mildest and IV the most severe form of PH. Number of participants per change in number of classes is reported.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 21
Participants
  -3 classes | 0
  -2 classes | 0
  -1 classes | 0
  0 classes | 21
  1 classes | 0
  2 classes | 0
  3 classes | 0

24. Secondary Outcome: Change in NT-proBNP From Baseline
Description: Laboratory biomarkers N-terminal prohormone brain-type natriuretic peptide (NT-proBNP) or brain-type natriuretic peptide (BNP) were tested for the participants. When both tests were available, NT-proBNP was chosen over BNP and the same test was performed at every required visit.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 14
picograms per milliliter (pg/mL) | -65.77 (585.41) [lower limit 585.41]

25. Secondary Outcome: Change in BNP From Baseline
Description: as for outcome 24
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 6
Picograms per milliliter (pg/mL) | 7.45 (10.65) [lower limit 10.65]

26. Secondary Outcome: Change in Quality of Life Evaluated by SF-10 Questionnaire From Baseline
Description: SF-10 is a parent-completed health survey for children that contains 10 questions adapted from the Child Health Questionnaire. It is scored using nom-based scoring to produce physical and psychosocial health summary measures. The possible range for the physical measure is -10.9 to 57.2 scores and the possible range for the psychosocial measure is 8.8 to 62.3 scores. Higher scores indicate more favorable functioning.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 21
Scores on a scale
  Physical summary score | 5.79 (12.46) [lower limit 12.46]
  Psychosocial summary score | 1.10 (6.85) [lower limit 6.85]

27. Secondary Outcome: Change in Quality of Life Evaluated by PedsQL Scale
Description: The PedsQL Generic Core Scales were designed to measure health-related quality of life in children and adolescents. It has 4 dimensions: physical functioning, emotional functioning, social functioning and school functioning. 3 Summary Scores of PedsQL were calculated from the scales including total scale score (23 questions), physical health summary score (physical functioning, 8 questions) and psychosocial health summary score (emotional, social and school functioning, 15 questions). Responses of the questions are transformed to a 0-100 scale. Higher scores indicate better quality of life.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 19
Scores on a scale
  Total scale score | 3.49 (10.81) [lower limit 10.81]
  Physical health summary score | 4.28 (13.51) [lower limit 13.51]
  Psychosocial health summary score | 3.07 (11.21) [lower limit 11.21]

28. Secondary Outcome: Number of Subjects With Clinical Worsening
Description: Clinical worsening was defined as: hospitalization for right heart failure, death, lung transplantation, Pott's anastomosis and atrioseptostomy, worsening of pulmonary arterial hypertension (PAH) symptoms, which must include either an increase in World Health Organization (WHO) functional class or appearance/worsening symptoms of right heart failure and need for additional PAH therapy.
Time Frame: Up to Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 24
Participants | 2

29. Secondary Outcome: Change in Estimated Right Atrial Pressure From Baseline
Description: Estimated right atrial pressure was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 16
millimetre of mercury (mmHg) | -0.6 (3.6) [lower limit 3.6]

30. Secondary Outcome: Change in Left Ventricular Eccentricity Index From Baseline
Description: Left ventricular (LV) eccentricity index (EI) was measured by echocardiography and defined as the ratio of the LV anteroposterior dimension to the septolateral dimension in the parasternal short-axis window by echocardiography. The value of EI greater than 1.0 is abnormal and suggests right ventricle (RV) overload.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 15
Ratio | 0.002 (0.907) [lower limit 0.907]

31. Secondary Outcome: Change in Pericardial Effusion From Baseline
Description: Pericardial effusion was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 1
Millimeter (mm) | 1.040 (NA) — Value was not calculated due to very low number of participants.

32. Secondary Outcome: Change in Pulmonary Artery Acceleration Time From Baseline
Description: Pulmonary artery acceleration time was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 15
Millisecond (msec) | -7.777 (35.898) [lower limit 35.898]

33. Secondary Outcome: Change in Right Ventricular Cardiac Index From Baseline
Description: Right ventricle (RV) cardiac index (CI) was measured by echocardiography and calculated by dividing the cardiac output (stroke volume × heart rate) by the body surface area. The change in RV CI should not be understood solely but associated with other conditions of the participants.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Liter/minute/square meter (L/min/m^2)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 13
Liter/minute/square meter (L/min/m^2) | 0.188 (2.094) [lower limit 2.094]

34. Secondary Outcome: Change in Right Ventricular Cardiac Output From Baseline
Description: Right ventricular cardiac output was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Liter per minute (L/min)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 13
Liter per minute (L/min) | 0.457 (3.066) [lower limit 3.066]

35. Secondary Outcome: Change in Right Atrial Diastolic Area From Baseline
Description: Right atrial diastolic area was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Square centimeter (cm^2)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 16
Square centimeter (cm^2) | 1.078 (3.330) [lower limit 3.330]

36. Secondary Outcome: Change in Right Atrial Diastolic Area Index From Baseline
Description: Right atrial (RA) diastolic area index was measured by echocardiography and calculated by dividing the RA area at end-diastole by the body surface area. The RA area index is a reflection of RA volume at end-diastole. The change in the index should not be understood solely but associated with other conditions of the participants.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 16
Ratio | 0.643 (2.314) [lower limit 2.314]

37. Secondary Outcome: Change in Right Atrial Systolic Area From Baseline
Description: Right atrial systolic area was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Square centimeter (cm^2)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 16
Square centimeter (cm^2) | 0.424 (3.758) [lower limit 3.758]

38. Secondary Outcome: Change in Right Atrial Systolic Area Index From Baseline
Description: Right atrial (RA) systolic area index was measured by echocardiography and calculated by dividing the RA area at end-systole by the body surface area. The RA area index is a reflection of RA volume at end-systole. The change in the index should not be understood solely but associated with other conditions of the participants.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 16
Ratio | 0.329 (2.417) [lower limit 2.417]

39. Secondary Outcome: Change in Right Ventricular Fractional Area Change From Baseline
Description: Right ventricular fractional area change was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Percentage (%) of area
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 15
Percentage (%) of area | -4.3 (7.3) [lower limit 7.3]

40. Secondary Outcome: Change in Right Ventricular Diastolic Area From Baseline
Description: Right ventricular diastolic area was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Square centimeter (cm^2)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 15
Square centimeter (cm^2) | 0.618 (4.519) [lower limit 4.519]

41. Secondary Outcome: Change in Right Ventricular Diastolic Area Index From Baseline
Description: Right ventricular (RV) diastolic area index was measured by echocardiography and calculated by dividing the RV area at end-diastole by the body surface area. The RV area index is a reflection of RV volume at end-diastole. The change in the index should not be understood solely but associated with other conditions of the participants.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 15
Ratio | 0.451 (3.562) [lower limit 3.562]

42. Secondary Outcome: Change in Right Ventricular Systolic Area From Baseline
Description: Right ventricular systolic area was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Square centimeter (cm^2)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 15
Square centimeter (cm^2) | 1.725 (3.847) [lower limit 3.847]

43. Secondary Outcome: Change in Right Ventricular Systolic Area Index From Baseline
Description: Right ventricular (RV) systolic area index was measured by echocardiography and calculated by dividing the RV area at end-systole by the body surface area. The RV area index is a reflection of RV volume at end-systole. The change in the index should not be understood solely but associated with other conditions of the participants.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 15
Ratio | 1.244 (3.277) [lower limit 3.277]

44. Secondary Outcome: Change in Systolic Pulmonary Artery Pressure From Baseline
Description: Systolic pulmonary artery pressure was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 3
millimetre of mercury (mmHg) | 5.7 (49.0) [lower limit 49.0]

45. Secondary Outcome: Change in Tricuspid Annular Plane Systolic Excursion From Baseline
Description: Tricuspid annular plane systolic excursion (TAPSE) was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 15
Millimeter (mm) | -1.27 (3.87) [lower limit 3.87]

46. Secondary Outcome: Change in Tricuspid Regurgitation Peak Velocity From Baseline
Description: Tricuspid regurgitation peak velocity was measured by echocardiography.
Time Frame: Baseline and Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Mean (Standard Deviation); unit: Meter/second (m/s)
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 10
Meter/second (m/s) | -0.085 (0.726) [lower limit 0.726]

47. Other Pre Specified Outcome: Taste and Texture (Questions 1 to 4) of the Oral Suspension of Riociguat at Week 0
Description: To assess the taste and texture of oral suspension of Riociguat, a questionnaire including 7 questions was used. Responses to Questions 1 to 4 are reported in this endpoint. Questions 1 and 2 were asked before the participants received the suspension; whereas questions 3 and 4 were asked right after administration of the suspension. Participants were asked to respond to the 4 questions as "yes" (= positive answer), "I do not know/unsure"(= indifferent answer) or "No" (= negative answer).
Time Frame: At the beginning of the treatment (Week 0)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 16
Participants
  Like the look of the drink: Yes | 4
  Like the look of the drink: No | 2
  Like the look of the drink: Unsure | 9
  Like the look of the drink: Missing | 1
  Like the smell of the drink: Yes | 4
  Like the smell of the drink: No | 2
  Like the smell of the drink: Unsure | 9
  Like the smell of the drink: Missing | 1
  Like the drink: Yes | 9
  Like the drink: No | 1
  Like the drink: Unsure | 5
  Like the drink: Missing | 1
  Like to drink again: Yes | 12
  Like to drink again: No | 0
  Like to drink again: Unsure | 3
  Like to drink again: Missing | 1

48. Other Pre Specified Outcome: Taste and Texture (Questions 1 to 4) the Oral Suspension of Riociguat at Week 24
Description: as for outcome 47
Time Frame: Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 14
Participants
  Like the look of the drink: Yes | 6
  Like the look of the drink: No | 1
  Like the look of the drink: Unsure | 6
  Like the look of the drink: Missing | 1
  Like the smell of the drink: Yes | 7
  Like the smell of the drink: No | 2
  Like the smell of the drink: Unsure | 4
  Like the smell of the drink: Missing | 1
  Like the drink: Yes | 6
  Like the drink: No | 4
  Like the drink: Unsure | 3
  Like the drink: Missing | 1
  Like to drink again: Yes | 6
  Like to drink again: No | 3
  Like to drink again: Unsure | 4
  Like to drink again: Missing | 1

49. Other Pre Specified Outcome: Taste and Texture (Question 5) of the Oral Suspension of Riociguat at Week 0
Description: To assess the taste and texture of oral suspension of Riociguat, a questionnaire including 7 questions was used. Number of participants per responses to Questions 5 "Taste of the drink" is reported in this endpoint. Question 5 was only asked to participants who answered "No" to Question 3 "Did you like the drink" or Question 4 "Would you like to drink this again". Participants were asked to answer "yes", "I do not know/unsure" or "No" to each taste including "sweet, sour, bitter, salty, disgusting and fruity".
Time Frame: At the beginning of the treatment (Week 0)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 1
Participants
  Sweet: Yes | 1
  Sweet: No | 0
  Sweet: Unsure | 0
  Sour: Yes | 0
  Sour: No | 1
  Sour: Unsure | 0
  Bitter: Yes | 0
  Bitter: No | 1
  Bitter: Unsure | 0
  Salty: Yes | 0
  Salty: No | 1
  Salty: Unsure | 0
  Disgusting: Yes | 0
  Disgusting: No | 1
  Disgusting: Unsure | 0
  Fruity: Yes | 1
  Fruity: No | 0
  Fruity: Unsure | 0

50. Other Pre Specified Outcome: Taste and Texture (Question 5) of the Oral Suspension of Riociguat at Week 24
Description: as for outcome 49
Time Frame: Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 4
Participants
  Sweet: Yes | 2
  Sweet: No | 1
  Sweet: Unsure | 1
  Sour: Yes | 1
  Sour: No | 3
  Sour: Unsure | 0
  Bitter: Yes | 0
  Bitter: No | 3
  Bitter: Unsure | 1
  Salty: Yes | 0
  Salty: No | 4
  Salty: Unsure | 0
  Disgusting: Yes | 4
  Disgusting: No | 0
  Disgusting: Unsure | 0
  Fruity: Yes | 0
  Fruity: No | 2
  Fruity: Unsure | 2

51. Other Pre Specified Outcome: Taste and Texture (Question 6) of the Oral Suspension of Riociguat at Week 0
Description: To assess the taste and texture of oral suspension of Riociguat, a questionnaire including 7 questions was used. Number of participants per responses to Questions 6 "Drink feels in mouth" is reported in this endpoint. Question 6 was only asked to participants who answered "No" to Question 3 "Did you like the drink" or Question 4 "Would you like to drink this again". Participants were asked to answer "yes", "I do not know/unsure" or "No" to each feeling including "like sand, sticky, gooey, slimy, creamy".
Time Frame: At the beginning of the treatment (Week 0)
Population: Participants in safety analysis set (SAF) with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 1
Participants
  Like Sand: Yes | 0
  Like Sand: No | 1
  Like Sand: Unsure | 0
  Sticky: Yes | 0
  Sticky: No | 1
  Sticky: Unsure | 0
  Gooey: Yes | 0
  Gooey: No | 1
  Gooey: Unsure | 0
  Slimy: Yes | 0
  Slimy: No | 1
  Slimy: Unsure | 0
  Creamy: Yes | 0
  Creamy: No | 1
  Creamy: Unsure | 0

52. Other Pre Specified Outcome: Taste and Texture (Question 6) of the Oral Suspension of Riociguat in Mouth at Week 24
Description: as for outcome 51
Time Frame: Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 4
Participants
  Like sand: Yes | 3
  Like sand: No | 1
  Like sand: Unsure | 0
  Sticky: Yes | 1
  Sticky: No | 3
  Sticky: Unsure | 0
  Gooey: Yes | 0
  Gooey: No | 3
  Gooey: Unsure | 1
  Slimy: Yes | 2
  Slimy: No | 1
  Slimy: Unsure | 1
  Creamy: Yes | 0
  Creamy: No | 2
  Creamy: Unsure | 2

53. Other Pre Specified Outcome: Taste and Texture (Question 7) of the Oral Suspension of Riociguat in Mouth at Week 0
Description: To assess the taste and texture of oral suspension of Riociguat, a questionnaire including 7 questions was used. Number of participants per responses to Questions 7 "Did you like the taste after swallowing" is reported in this endpoint. Question 7 was only asked to participants who answered "No" to Question 3 "Did you like the drink" or Question 4 "Would you like to drink this again". Participants were asked to respond as "yes" (= positive answer), "I do not know/unsure"(= indifferent answer) or "No" (= negative answer).
Time Frame: At the beginning of the treatment (Week 0)
Population: Participants in safety analysis set (SAF) with assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 1
Participants
  Like the taste after swallowing - Yes | 1
  Like the taste after swallowing - No | 0
  Like the taste after swallowing - Unsure | 0

54. Other Pre Specified Outcome: Taste and Texture (Question 7) of the Oral Suspension of Riociguat in Mouth at Week 24
Description: as for outcome 53
Time Frame: Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 4
Participants
  Like the taste after swallowing - Yes | 0
  Like the taste after swallowing - No | 3
  Like the taste after swallowing - Unsure | 1

55. Other Pre Specified Outcome: Expression Assessment on the Taste and Texture of Oral Suspension of Riociguat - Week 0
Description: The facial expression of the subjects concerning appearance, smell and taste of the suspension of Riociguat was captured by the investigators as "comfortable", "indifferent" and "displeased".
Time Frame: At the beginning of the treatment (Week 0)
Population: Participants in safety analysis set (SAF) with assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 16
Participants
  Comfortable | 7
  Indifferent | 8
  Displeased | 0
  Missing | 1

56. Other Pre Specified Outcome: Expression Assessment on the Taste and Texture of Oral Suspension of Riociguat - Week 24
Description: as for outcome 55
Time Frame: Week 24 (plus/minus 5 days)
Population: Participants in safety analysis set (SAF) with assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat >=6 to <18 Years
Number analyzed (Participants) | 14
Participants
  Comfortable | 6
  Indifferent | 5
  Displeased | 2
  Missing | 1

ADVERSE EVENTS:
Time Frame: From start of study drug up to 2 days after the last dose of study drug in the main study part, up to 24 weeks plus/minus 5 days.
Arm/Group | Riociguat >=6 to <18 Years
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 4/24
Other Adverse Events (participants affected / at risk) | 15/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat >=6 to <18 Years (N=24)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 2 (2)
Vascular device infection (Infections and infestations) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat >=6 to <18 Years (N=24)
Pyrexia (General disorders) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (7)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 7 (11)
Hypotension (Vascular disorders) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (5)

LIMITATIONS AND CAVEATS:
The results should be interpreted with caution due to the limited number of subjects. The number of subjects with clinical worsening events was too low to produce valid Kaplan-Meier estimates for the time to clinical worsening.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Most restricted agreement: CTA Japan; Embargo time mentioned. Hospital shall obtain prior written consent of Sponsor if PI intends to publish the information obtained from study externally such as in a professional society or association.

DOCUMENTS (2):
  • Study Protocol (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT02562235/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT02562235/SAP_001.pdf